CLINICAL TRIAL: NCT03670719
Title: Effectiveness of Manual Therapy and Exercise vs Exercise in Subjects With Chronic Cervical Pain and Upper Cervical Spine Dysfunction: A Randomized Controlled Trial
Brief Title: Effectiveness of Manual Therapy and Exercise vs Exercise in Subjects With Chronic Cervical Pain and Upper Cervical Spine Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez-Sanz, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N13/2018
Record Dates: First submitted 2018-09-06; First posted 2018-09-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Neck Pain; Cervical Pain
Keywords: manual therapy; exercise; physiotherapy; chronic cervical pain; upper cervical spain
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the evaluator is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy and Exercise Group (Experimental): Combination of manual therapy and exercises for chronic cervical pain
  Interventions: Other: Manual Therapy and Exercise
- Exercise Group (Active Comparator): Only exercises for chronic cervical pain
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Manual Therapy and Exercise — Combination of physiotherapy (manual therapy) techniques and exercises for the cervical spine
  Arms: Manual Therapy and Exercise Group
Other: Exercise — Exercises for the cervical spine
  Arms: Exercise Group

SUMMARY:
There is a lot of scientific evidence about the effectiveness of manual therapy and exercise / training in subjects with cervical pain. Most of the high quality systematic reviews agree on the need to combine manual therapy and exercise for the treatment of chronic cervical pain. However, articles that focus on manual therapy in the treatment of the upper cervical spine are not as common, being that the most commonly prescribed exercises are those of craniocervical flexion, (flexion of the upper cervical spine).

The investigators believe that participants who are going to benefit more from the integration of manual therapy and exercise will be those who have a real restriction of the upper cervical spine, and for these, is indispensable, the application of manual therapy techniques before the integration of the active exercise to obtain optimal results.

This project is going to try to define participants with chronic cervical pain and upper cervical spine restriction that may benefit more from the combination of manual therapy and exercise than the rest. The investigators are going to study changes in different variables about function, pain, ultrasound, muscle tone, joints... Strengthen the importance of specificity in physiotherapy interventions and increase the evidence on the importance of manual therapy in a subgroup of participants with chronic cervical pain, improve knowledge about the involvement of the upper cervical spine in cervical pathology and check the effectiveness of a self-treatment program for participants with chronic cervical pain.

The objective of this trial is to compare the effectiveness of an integrative approach of manual therapy associated with exercise versus exercise in participants with chronic cervical pain and upper cervical spine dysfunction.

For this purpose, the investigators conduct a randomized controlled trial, simple-blind (Only is possible to blind the evaluator).

The Sample size is 52 participants (2 groups of 26 participants). One of the groups will receive 4 training sessions with exercises for the cervical spine between 30 and 45 minutes duration per session and the other group will receive 4 sessions of a combination of manual therapy and training exercises also between 30 and 45 minutes each session. In addition, all participants will receive self-treatment techniques for self-management of their dysfunction.

Cervical exercises will consist of a set of training techniques to improve the function and symptomatology that the participant has. These exercises have been widely evidenced and do not suppose any health risk.

The techniques of manual therapy can be the manipulation technique in resting position, vertebral mobilization and / or musculature (massage and / or stretching). All the treatments applied follow the safety recommendations of the International Federation of Orthopedic Manual Therapists (IFOMPT). If participants need clarification, they can talk to the principal investigator (Jacobo Rodríguez Sanz) at any time.

One physiotherapist will perform the physical examination, and a different one will apply the treatment. Physical therapists doing the screening will not know which group has been assigned to them, so the participant will be asked not to provide the evaluators any information about the assignment of his group to improve the quality of the study.

The examination will consist of tests to assess whether the participant is a candidate to participate in the study, the measurement of pain, the exhaustive assessment of all cervical musculature with different measuring instruments and the measurement of joint mobility.

The first day theparticipant be given information about his pain, his daily habits and activities that he usually does.

The assessment of his problem will consist in the measurement of the amount of movement he can makes in the cervical area without pain, the ability to orient himself in certain movements with his eyes closed, the intensity of his pain, the evaluation of the state of his muscles. stabilizing as a mobilizer through ultrasound, muscle test and palpation. The functionality of his cervical vertebrae will also be evaluated and he will be asked different questionnaires about the functionality, pain and condition of his cervical pain, headache (in case of suffering) and kinesiophobia.

Both the evaluation and the treatment will be without pain. In addition, he will be given a series of personalized exercises to improve his problem, which must be done every day during the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Medical diagnosis of chronic cervical pain (more than 3 months of cervical pain evolution)
* Positive flexion rotation test

Exclusion Criteria:

* Recent spine, head or mouth surgery.
* Diabetes mellitus
* Recent infection and/or inflammatory arthritis, and cervical and/or brain traumatism records.
* Contraindication for manual therapy or cervical training

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index (NDI) Questionnaire | Change between baseline (immediately before intervention) and post intervention (1 month), after 3 months
  The NDI is a modification of the Oswestry Low Back Pain Disability Index . It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain
Change in Flexion Rotation Test (FRT) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention), and post intervention (1 month) after 3 months
  This test is used to see the amount of movement of the upper cervical spine and is the test most used in the literature. It is positive when there is a decrease of 10 degrees or more in the cervical rotation with maximum flexion, in a sense with respect to the contralateral or presents hypomobility of segment C1 with a mobility less than 32º

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold | Change between baseline(immediately before intervention) and post intervention (immediately after intervention), and post intervention (1 month) after 3 months
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom. This force is applied by a portable and digital machine. This machine has a push button so the patient can press at the moment in which the applied force begins to be slightly painful. When the patient presses the button, the evaluator registers the number that appears on the screen.
Change in Cervical Range of Movement | Change between baseline(immediately before intervention) and post intervention (immediately after intervention), and post intervention (1 month), after 3 months
Change in Numeric Pain Rating Scale (NPRS) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention), and post intervention (1 month), after 3 months
  The Numeric Pain Rating Scale (NPRS) is a one-dimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes.
Change in Ultrasound | Change between baseline(immediately before intervention) and post intervention (1 month), after 3 months
  To measure the thickness of the longus colli muscle

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Rodríguez-Sanz, Pt, Principal Investigator — Physiotherapy Research Unit, University of Zaragoza
Locations (1):
- Faculty of Health Sciences of University of Zaragoza, Zaragoza, Spain